CLINICAL TRIAL: NCT05344794
Title: Relationship Between Serum N/OFQ and Cerebral Cardiac Syndrome After Stroke
Brief Title: Relationship Between Serum N/OFQ and Brain-heart Syndrome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zheng Guo (Other)
Responsible Party: Sponsor-Investigator, Zheng Guo, professor, Second Hospital of Shanxi Medical University
Organization: Second Hospital of Shanxi Medical University (Other)
Other Study IDs: hanyi20220418
Record Dates: First submitted 2022-04-18; First posted 2022-04-25 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Cerebral-Cardiac Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CCS group: Patients with cerebral syndrome diagnosed by the Second Hospital of Shanxi Medical University
  Interventions: Diagnostic Test: Enzyme-linked immunosorbent assay
- Control group: Patients who have not had a cerebral syndrome in ischemic stroke
  Interventions: Diagnostic Test: Enzyme-linked immunosorbent assay

INTERVENTIONS:
Diagnostic Test: Enzyme-linked immunosorbent assay — Serum N/OFQ , IL-6 and NE levels were detected.

SUMMARY:
Choosing the neurology patients in the Second Hospital of Shanxi Medical University, diagnosed with patients with cerebral syndrome into the experimental group; patients who did not have cerebral syndrome included in the control group, and all selected people had no intimate relationship with each other.Specimen collecting control group and the study group serum inflammatory factor IL-6, solvent peptide and catecholamine content. The difference between the two groups of data was observed.According to the literature, it is guess: The solitary peptide content of the experimental group will be higher than the control group, and is positively correlated with IL-6, catecholamine content.The difference was statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic criteria in compliance with cerebral syndrome
* Acute ischemic stroke patients in line with the "Chinese Acute Ischemic Stroke Treatment Guide 2018" related diagnostic criteria
* There is no intimate relationship between all selected people and knows this study, and signs informed consent

Exclusion Criteria:

* Heart-type cerebral infarction, hemorrhagic stroke, brain tumor and past intracranial hemorrhage
* Complicated with severe cardiovascular complications (such as coronary heart disease, acute coronary syndrome, acute myocardial infarction, chronic heart failure, atrial fibrillation, etc.)
* Complicated with severe liver and kidney dysfunction (such as coagulous dysfunction, cirrhosis, nephrotic syndrome , Renal failure, etc.)
* Complicated with severe diabetes complications (such as diabetic nephropathy, diabetic foot, diabetic acidosis, high blood sugar hypertonic state, diabetes coronary heart disease, etc.)
* Complicated with Psychological disease
* Complicated with chronic obstructive pulmonary disease(COPD)
* BMI> 40

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in the Second Hospital of Shanxi Medical University from May 2022 to October 2023
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-10-31 (Estimated)

PRIMARY OUTCOMES:
N/OFQ | 24 hours
  Serum N/OFQ levels
IL-6 | 24 hours
  Serum IL-6 levels
NE | 24 hours
  Serum NE levels

CONTACTS AND LOCATIONS:
Locations (1):
- Second of Shanxi Medical University, Taiyuan, Shanxi, China